CLINICAL TRIAL: NCT04619524
Title: Biomarkers of Endometrial Receptivity: A Prospective Multicenter Study on Proteomic Biomarkers of Endometrial Receptivity in Cervical Mucus ( PRO BIOMER - CM )
Brief Title: Biomarkers of Endometrial Receptivity
Acronym: BIOMER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Institute of Molecular and Translational Medicine, Czech Republic (Other)
Collaborators: University Hospital Olomouc (Other); Brno University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4616-27870
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: IVF; Infertility Treatment; Fertility Disorders; Embryo Transfer
Keywords: cervix; mucus; endometrium; receptivity; biomarker; proteomics; infertility; in-vitro; fertilisation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Patients undergo cycle with the transfer of fresh embryos (Experimental): In study group A the cervical mucus will be collected from patients undergoing the in vitro fertilisation (IVF)/intracytoplasmic sperm injection (ICSI)/embryo transfer (ET) cycle with the transfer of fresh embryos.
  Interventions: Diagnostic Test: Cervical mucus will be collected from patients undergoing IVF
- B: Patients undergo cycle with the transfer of frozen embryos (Experimental): In study group B cervical mucus will be sampled from patients undergoing treatment cycles with the transfer of cryopreserved embryos.
  Interventions: Diagnostic Test: Cervical mucus will be collected from patients undergoing transfer of cryopreserved embryos

INTERVENTIONS:
Diagnostic Test: Cervical mucus will be collected from patients undergoing IVF — Patients undergoing hormonal stimulation for IVF will be sampled for cervical mucus.
  Arms: A: Patients undergo cycle with the transfer of fresh embryos
Diagnostic Test: Cervical mucus will be collected from patients undergoing transfer of cryopreserved embryos — Patients undergoing hormonal substitution for transfer of cryopreserved embryos will be sampled for cervical mucus.
  Arms: B: Patients undergo cycle with the transfer of frozen embryos

SUMMARY:
Analysis of proteins from cervical mucus will be done in patients undergoing infertility treatment (fresh or frozen embryo transfer). Cervical mucus will be analysed for potential new biomarkers of endometrium receptivity. Comparison of the peptide spectrum will be done for the pregnant and not pregnant patients.

DETAILED DESCRIPTION:
Successful implantation depends on synchronization between a normal functional embryo at the blastocyst developmental stage and a receptive endometrium. The endometrium is receptive to blastocysts during a spatially and temporally restricted time window called the "window of implantation". Failure of the endometrium to attain receptivity is one cause of infertility, and this is not currently assessed during infertility workup due to a lack of reliable markers for receptivity. Better tests are required to assist the clinician with the decision when to defer a transfer and to freeze all embryos. Proteomics, or the analysis of the proteins in any sample, provides physiologically relevant information, since there are many regulatory steps between the transcriptome and functional proteins. Uterine fluid is a protein-rich histotroph that contains, among other components, secretions from the endometrial glands and cleavage products of both the secreted proteins and the glycocalyx. The aim of this study is to assess the highly sensitive mass spectrometer analysis of the proteins from cervical mucus for the detection of defects in endometrial receptivity and search for new endometrial receptivity biomarkers.

ELIGIBILITY:
Inclusion Criteria - Arm A - stimulated cycle:

* female aged less than 37 years (maximally 36y + 364d)
* no smoker
* normal menstrual cycles lasting between 25 to 35 days
* had been infertile for less than five years
* normal responder
* fewer than three failed cycles of assisted reproduction treatment, including fresh IVF/ intracytoplasmic sperm injection (ICSI) embryo transfer cycles and/or frozen-thawed embryo transfer cycles
* sperm obtained through ejaculation
* spermiogram more than 5 million sperm/mL
* BMI 19-29 kg/m2
* follicle stimulating hormone (FSH) < 10 IU/L on the third day
* basal antral follicle count of 5-15
* undergoing the same routine gonadotrophin-releasing hormone agonist (GnRHa) long depot or gonadotrophin-releasing hormone antagonist (GnRH-ant.) protocol
* informed consent

Exclusion Criteria - Arm A - stimulated cycle:

* genetic disease
* metabolic and/or endocrine disorders
* polycystic ovary syndrome (defined by the Rotterdam criteria)
* women with prior diagnosis of endometriosis or adenomyosis
* previous gynecological/pelvic surgery except for salpingectomy
* repeated spontaneous abortions (two or more)
* previously less than 5 oocytes and/or serum anti-Mullerian hormone value < 1.0 mIU/ml or more than 20 oocytes, milli-International unit (mIU)
* previous ovarian hyperstimulation syndrome (OHSS)
* presence of any structural abnormality of the reproductive system
* donor oocyte cycles
* severe male factor infertility < 5 million sperm/mL
* low response to stimulation
* endometrium < 8 mm at the day of human chorionic gonadotropin (hCG) or ET
* number of retrieved oocytes 5 - 20
* low fertilization capacity (rate of fertilization < 20% and late ICSI following IVF fertilization failure)
* OHSS
* IVF cycle cancelled before ET
* other than easy one high-quality blastocyst transfer (at least grade 3BB)

Inclusion criteria - Arm B - substituted cycle:

* female aged less than 37 years (maximally 36y + 364d)
* no smoker
* normal menstrual cycles lasting between 25 to 35 days
* had been infertile for less than five years
* normal responder at stimulation
* fewer than three failed cycles of assisted reproduction treatment, including fresh IVF/ intracytoplasmic sperm injection (ICSI) embryo transfer cycles and/or frozen-thawed embryo transfer cycles
* sperm obtained through ejaculation
* spermiogram more than 5 million sperm/mL
* BMI 19-29 kg/m2
* FSH < 10 IU/L on the third day
* undergoing the same routine estrogen/progesterone substituted cycle
* informed consent

Exclusion criteria - Arm B - substituted cycle:

* genetic disease
* metabolic and/or endocrine disorders such as diabetes, metabolic syndrome, and thyroid disorders
* polycystic ovary syndrome (defined by the Rotterdam criteria), hyperprolactinaemia
* women with prior diagnosis of endometriosis or adenomyosis
* previous gynecological/pelvic surgery except for salpingectomy
* repeated spontaneous abortions (two or more)
* previously less than 5 oocytes and/or serum anti-Mullerian hormone value < 0.5 mIU/ml in the stimulated cycle
* previous OHSS
* presence of any structural abnormality of the reproductive system
* severe male factor infertility < 5 million sperm/mL in the stimulated cycle
* number of retrieved oocytes 5 - 20 in the stimulated cycle
* low fertilization capacity (rate of fertilization < 20% and late ICSI following IVF fertilization failure)
* endometrium less than 8 mm at the day of thawing and transfer indication
* thawed blastocyst cycle cancelled before ET
* other than easy one best quality frozen/thawed blastocyst transfer (at least grade 3BB)

Max Age: 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 476 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mass spectrometer analysis of the proteins from cervical mucus | 48 months
  Highly sensitive mass analysis of the proteins from cervical mucus on Thermo Orbitrap Elite instrument for all collected samples.

SECONDARY OUTCOMES:
Comparison of the protein analysis between the pregnant and not pregnant patients | 48 months
  Comparison of the protein analysis (qualitative and quantitative) will be done between the pregnant and not pregnant patients. Pregnant patients will be followed-up until child delivery.
Detection of the new endometrial receptivity biomarkers. | 48 months
  Proteomic endometrial receptivity biomarkers will be detected based on the analysis of measured data in relation to the successful implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Marian Hajduch, MD.PhD., Study Director — Palacky University in Olomouc, Faculty of Medicine and Dentristry
Locations (2):
- Czechia (2):
  - Brno University Hospital, Brno, South Moravian
  - University Hospital Olomouc, Olomouc